CLINICAL TRIAL: NCT01544387
Title: PPROM: Bed Rest Versus Activity Trial (BRAT)
Brief Title: Preterm Premature Rupture of Membranes (PPROM): Bed Rest Versus Activity Trial
Acronym: BRAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 10-0352
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Pregnancy; Pre-term Premature Rupture of Membranes
Keywords: Preterm Premature Rupture Of Membranes; PPROM; Pregnancy; Bed rest.
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Bed Rest; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bed Rest (Other): Subjects will have limited activity. Bed Rest
  Interventions: Other: Bed Rest
- Activity (Other): Activity
  Interventions: Other: Activity

INTERVENTIONS:
Other: Bed Rest — * Subjects are admitted to their labor and delivery room and will spend the majority of their day in their hospital bed, usually in a reclined or sleeping position
  * Subjects will be instructed to refrain from walking or engaging in any extraneous activity, including lifting or spending any extended period of time out of bed
  * Subjects may have limited bathroom privileges
  Arms: Bed Rest
Other: Activity — * Subjects are admitted to their labor and delivery room and will spend the majority of their time in their hospital bed
  * Subjects will be given the opportunity of 3 periods of walking around their room and/or the hall on labor and delivery each day, each period consisting of approximately 20 minutes - this is the minimum activity level required for the study. Subjects are permitted more activity as desired.
  Arms: Activity

SUMMARY:
The objective of this study is to determine, through a randomized clinical trial, whether bed rest is helpful for the management of pregnancies complicated by preterm premature rupture of membranes (PPROM).

DETAILED DESCRIPTION:
Bed rest at home or in the hospital has been widely advised for many complications of pregnancy, including preterm premature rupture of membranes (PPROM) - a problem in which the water breaks prematurely and is not accompanied by labor. For most patients, bed rest represents a significant change in lifestyle, including having to stop work, and/or not being able to do household duties or take care of their children. In pregnancies, complicated by PPROM, patients are usually hospitalized and placed on bed rest throughout the stay.

Despite its widespread use, there are no good published studies evaluating the effect of bed rest on common complications of pregnancy. There are, on the other hand, several other studies that indicate that bed rest may actually be harmful. Bed rest has been shown to increase a patient's risk for developing blood clots in their legs or in their lungs. Bed rest may also have myriad other deleterious effects such as muscle and bone atrophy. Furthermore, bed rest has been shown to be emotionally distressing both to the patient and her family.

Once the amniotic membranes are broken, amniotic fluid will generally continue to leak for the remainder of the pregnancy, and a fetus in otherwise good health will continue to make more amniotic fluid by urination. In patients hospitalized with PPROM, an objective assessment that can be obtained is an ultrasound amniotic fluid index (AFI), which measures how much amniotic fluid remains despite the water having broken. It is thought that a greater amount of amniotic fluid may be indicative of a longer duration/continuation of pregnancy and fewer adverse interim effects such as cord compression. Remaining on bed rest was thought to perhaps affect the AFI in a positive way. It is unclear whether retaining the ability to ambulate would affect the AFI, because amniotic fluid continues to leak even while on bed rest; the benefits of ambulation may be well worthwhile. Twice weekly ultrasound amniotic fluid measurement will be checked to assess the effects of ambulation verses bed rest in pregnancies complicated by PPROM, and secondarily look at the overall outcome of the pregnancy.

The objective of this study is to determine, through a randomized clinical trial, whether bed rest is helpful for the management of pregnancies complicated by preterm premature rupture of membranes.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria
* Pregnant women
* Clinical diagnosis of PPROM (made by sterile speculum examination)
* Singleton pregnancy
* Vertex or frank breech presentation
* 18-55 years old
* Gestational age < 34 weeks

Exclusion Criteria:

* Multiple gestations
* Gestational age > 34 weeks
* Current treatment with MgSO4 for preterm labor
* Footling breech presentation
* Any maternal or fetal indication for immediate delivery

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
AFI | From admission to delivery, average 6-7 days
  primary outcome is the amniotic fluid index (AFI) - a 4 quadrant measurement of the amniotic fluid surrounding the fetus.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Stone, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Elmhurst Hospital Center, Elmhurst, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Bigelow CA, Factor SH, Miller M, Weintraub A, Stone J. Pilot Randomized Controlled Trial to Evaluate the Impact of Bed Rest on Maternal and Fetal Outcomes in Women with Preterm Premature Rupture of the Membranes. Am J Perinatol. 2016 Mar;33(4):356-63. doi: 10.1055/s-0035-1564427. Epub 2015 Oct 13. PMID 26461925